CLINICAL TRIAL: NCT05302310
Title: INSPIRE: Feasibility of a Community-based Integrated Care Model for Older Adults Living at Home
Acronym: INSPIRE
Status: Completed | Type: Observational
Sponsor: University of Basel (Other)
Collaborators: Swiss Tropical & Public Health Institute (Other); Basel Institute for Clinical Epidemiology and Biostatistics (Other); KU Leuven (Other); Aerztegesellschaft Basellland (Unknown); University of Zurich (Other); Duke University (Other); Swiss National Science Foundation (Other); Basel-Landschaft Swisslos (Unknown); European Commission (Other); Basel-Landschaft volkswirtschafts- und gesundheitsdirektion (Unknown)
Responsible Party: Principal Investigator, Sabina De Geest, Prof. Dr., University of Basel
Other Study IDs: INSPIRE Feasibility study
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Frailty
Keywords: Feasibility; Delivery of Health Care, Integrated; implementation science; advance practice nurse
MeSH Terms: conditions — Frailty | interventions — Delivery of Health Care, Integrated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (6):
- Older adults (1A): All older adults visiting/contacting the Information and Advice Center
- Older adults (1B): These older adults will receive the integrated care (intervention) provided by the nurse and the social worker of the Information and Advice Center
  Interventions: Other: integrated care
- Older adults (1C): This group corresponds to a nested sample of older adults who will receive the integrated care (intervention) provided by the nurse and the social worker of the Information and Advice Center and will participate in interviews with the research team.
  Interventions: Other: integrated care
- Informal caregivers (2): The informal caregivers of older adults receiving the integrated care (intervention) provided by the nurse and the social worker of the Information and Advice Center will participate in interviews with the research team.
- IAC nurse and social worker (3): The nurse and the social worker who provide the integrated care (intervention) in the Information and Advice Center will participate in bi-weekly meetings with the research team
- External collaborators (4): The external collaborators who are involved in the care of the participating older adults and have collaborated with the nurse and the social worker of the Information and Advice Center will complete a survey sent by mail or e-mail.

INTERVENTIONS:
Other: integrated care — i) Screening of older people for risk of frailty using a frailty screening tool, to identify the appropriate care they will require:
  * Older adults with low risk of frailty will receive health promotion and preventive care from the Information and Advice Center nurse and/or social worker.
  * Older adults at risk will receive the following:
  ii) a Comprehensive Geriatric Assessment (CGA) delivered by the Information and Advice Center nurse and social worker over the course of multiple appointments, to identify the health and social care needs and goals of the older person; iii) Development of an individualized care plan by a multidisciplinary team, which will include evidence-based interventions and be coordinated by the Information and Advice Center nurse and/or the social worker; and iv) follow-up depending on the situation of each older person, and adaptation of the individualized care plan, as needed.
  Groups: Older adults (1B); Older adults (1C)

SUMMARY:
Background: The care of older people, often suffering from multiple chronic health problems is complex. As a result, many home-dwelling older people receive long-term care by a large number of care providers often in various care settings, which are neither centralized nor coordinated, putting older people are at risk for fragmented care. To address the complex needs and overcome fragmentation of care, implementation of integrated care models has been recommended. Integrated care has been described as a person-centred model of care that is structured to support coordinated, pro-active care led by a multidisciplinary core team and a lead coordinator communicating and cooperating across and within health and social sectors. However, a systematic review and meta analysis published by our research team could not show convincing evidence regarding the beneficial impact of integrated care models on health and service outcomes. But our study highlighted that the majority of the studies included effectiveness outcomes only and lacked process and implementation outcomes hindering to determine whether the negative conclusions were due to intervention or implementation failure. Therefore, this indicates the need for effectiveness studies which include process evaluations, contextual analysis, and measuring proximal implementation outcomes to determine if, how and why community-based integrated care for frail older adults is successful in practice.

To facilitate the uptake of integrated care in daily practice and overcome implementation issues, principles and methods from the field of implementation science should be incorporated into future research.

In January 2018, the Canton Basel-Landschaft (BL) published a new legal framework to redesign care for home-dwelling older people in the canton. This legal framework mandates the reorganization of the Canton BL into larger care regions and the creation of an Information and Advice Center (IAC) in each of these care regions. The legislation mandates the IAC to be staffed with at least a nurse. Subsequently, the INSPIRE research team has been working together with the Canton and the care region of Leimental to help operationalize and evaluate a care model for the IAC.

The overall INSPIRE project is a three-phase implementation science project which aims to develop, implement and evaluate an integrated care model for the IAC for home-dwelling older adults in Canton BL. Phase 1: consisted in the development of the community-based integrated care model. Phase 2: We will assess the feasibility of the community-based integrated model of care at the IAC in Leimental. Phase 3: we will evaluate the effectiveness of this intervention.

The current study focuses in the phase 2.

Aims:

1. assess feasibility of recruitment to the IAC including external (e.g., strategies used to promote the IAC services) and internal processes (e.g., the number of visitors to the IAC; how clients heard of the IAC; among others);
2. assess the adoption, acceptability, feasibility, and fidelity of the integrated care model at the IAC BPA in Leimental;
3. explore perceptions of older adults and their caregivers, IAC staff, and external health and social care providers towards the implemented care model, and if adaptations are needed to the care model or the implementation strategies/process.

Design: The feasibility study uses multiple methods. For aim 1, a descriptive study will be conducted to monitor the strategies used to promote the IAC and to assess which ones worked in getting older adults to reach out to the IAC. To address aims 2 and 3, a parallel convergent mixed methods observational design will be used, being the core aspect of this phase. A combination of administrative data, health record reviews, older adult and informal caregiver interviews, IAC staff meetings, and a questionnaire of community professional collaborators will be used to meet the aims of the feasibility study.

Sample: For this study, multiple samples will be included to collect administrative data, implementation outcomes, and individual characteristics of consenting older adults who used the IAC services: external (people respondents to promotion strategies) and internal (all visitors to the IAC); older adults; frail older adults who receive a CGA and their informal caregivers; the IAC nurse and social worker; and community professionals who collaborate with the IAC in care coordination.

Measurements & Outcomes: Engagement measures will be provided by the IAC Administration about all visitors to the IAC. Implementation outcomes will be captured from IAC staff; older adults visiting the IAC (or with home appointments) and their informal caregivers; and community healthcare collaborators using a combination of meeting logs, interviews, IAC health records, and a questionnaire. The estimation of time-driven activity-based cost will be captured by using information provided by the IAC staff.

DETAILED DESCRIPTION:
Background The care of older people, often suffering from multiple chronic health problems is complex. As a result, many home-dwelling older people receive long-term care by a large number of care providers often in various care settings, which are neither centralized nor coordinated, putting older people are at risk for fragmented care. To address the complex needs and overcome fragmentation of care, implementation of integrated care models has been recommended. Integrated care has been described as a person-centred model of care that is structured to support coordinated, pro-active care led by a multidisciplinary core team and a lead coordinator communicating and cooperating across and within health and social sectors. However, a systematic review and meta analysis published by our research team could not show convincing evidence regarding the beneficial impact of integrated care models on health and service outcomes. But our study highlighted that the majority of the studies included effectiveness outcomes only and lacked process and implementation outcomes hindering to determine whether the negative conclusions were due to intervention or implementation failure. Therefore, this indicates the need for effectiveness studies which include process evaluations, contextual analysis, and measuring proximal implementation outcomes to determine if, how and why community-based integrated care for frail older adults is successful in practice.

To facilitate the uptake of integrated care in daily practice and overcome implementation issues, principles and methods from the field of implementation science should be incorporated into future research.

In January 2018, the Canton Basel-Landschaft (BL) published a new legal framework to redesign care for home-dwelling older people in the canton. This legal framework mandates the reorganization of the Canton BL into larger care regions and the creation of an Information and Advice Center (IAC) in each of these care regions. The legislation mandates the IAC to be staffed with at least a nurse. Subsequently, the INSPIRE research team has been working together with the Canton and the care region of Leimental to help operationalize and evaluate a care model for the IAC.

The overall INSPIRE project is a three-phase implementation science project which aims to develop, implement and evaluate an integrated care model for the IAC for home-dwelling older adults in Canton BL. Phase 1: We developed a community-based integrated care model. Phase 2: We will assess the feasibility of the community-based integrated model of care at the IAC in Leimental. Phase 3: we will evaluate the effectiveness of this intervention.

The current study focuses in the phase 2.

Hypothesis and primary objective

The primary objective of this feasibility study is to 1) assess feasibility of recruitment to the IAC and evaluate recruitment strategies 2) assess the adoption, acceptability, feasibility, and fidelity of the integrated care model at the IAC, and 3) explore perceptions of older adults and their caregivers, IAC staff, and health and social care providers (e.g., GP, Spitex Nurse) towards the implemented care model, and if adaptations are needed to the care model or the implementation strategies.

Project design

The feasibility study will be conducted in March 2022, using multiple methods. For objective 1, a descriptive study will be conducted to monitor the strategies used to promote the IAC and to assess which ones were effective. To address objectives 2 and 3, which are the core aspects of this study phase, a parallel convergent mixed methods observational design will be used (whereby both quantitative and qualitative data are collected during a similar time period, analyzed separately, then merged). The quantitative data sources will include: IAC administrative data, IAC health records, and the NoMAD survey, while qualitative sources will include: interviews and meeting logs. The study will take place in a single center (i.e., the IAC in the Leimental care region). Effectiveness outcomes are not within the scope of this study phase.

Screening and recruitment

Objective 1: external processes, including IAC outreach, are not conducted by the researchers. For internal processes, all IAC visitors (sample 1A) will be included in our sample. Recruitment-related data will by aggregated and sent to the INSPIRE research team by the IAC administrative staff, hence no recruitment/screening is needed.

Objectives 2 & 3: Older adults [sample 1B & 1C] and relatives/legal representatives

Recruitment will be done following these steps:

(i) Older adults' arriving at the IAC/receiving an appointment at their home, will be asked to fill in client information forms as part of his/her IAC health record, including the GFI screening tool (self-administered). The GFI score will help the nurse(s) to determine whether the older adult needs:

1. GFI < 4 = health promotion and prevention (no CGA); or
2. GFI ≥ 4 = full CGA The GFI score will therefore also determine whether the INSPIRE research team will invite the older adult for an interview.

(ii) For home-based older adults aged 64+ who have a health record created (sample 1B), the IAC nurse will inform them about the study and provide the INSPIRE study invitation letter (offering to read the letter for older adults depending on their preference. The nurse will ask if they are interested and agree for their contact information to be passed to the INSPIRE team. On a weekly basis, the INSPIRE team will reach out to the Nurse to identify potential participants for a IAC health record review (based on inclusion/exclusion criteria).

(iii) The research team representative will then reach out to confirm the invitation to the older adult and ask for consent for participation. The INSPIRE research team will either approach the older adult in the IAC, their home or by phone to explain the study procedures and ask for consent to review their IAC health record and to potentially participate in an interview. Consent will be documented by signature. After review of the IAC health record, only eligible older adults (e.g., aged 75+, CGA completed, GFI≥4; Sample 1C) will be contacted again to arrange an interview.

Proxy consent, if required: The nurse will assess cognition as part of the regular standard of care during the CGA. If the nurse is concerned about the older adults' capacity to consent to the research study based on the Mini-Cog assessment and their clinical judgement, a proxy consent will be sought (i.e., legal representative). In this case, when the nurse introduces the study to the older adult, he/she will also ask if the INSPIRE research team can reach out to their legal representative as well.

The INSPIRE research team will speak to the family member/legal representative and older adult, and will ask for proxy consent. If a proxy has consented for the interview, the interview can also be in presence of the proxy. If the proxy provides consent for the health record review but not for the interview (or if the individual does not want to complete an interview), the proxy will still be invited to complete the interview designed for informal caregivers.

Informal caregiver [sample 2] If an informal caregiver (e.g., family member or neighbour) attended the IAC appointment with an older adult, the older adult will be asked if we could also interview the informal caregiver to gather their perspective on the older adults' experience with the IAC. Given the crucial role informal caregivers play in the care and support of frail older adults who are living at home, it is beneficial to gather the informal caregivers' perspective of the feasibility and acceptability of the IAC appointments and if there were any barriers to participation. If the older adult agrees to an informal caregiver being contacted, the INSPIRE team will contact the informal caregiver to discuss the study procedures, the consent form, and arrange a time for the interview. The consent of the informal caregiver may be by signature, depending on the caregivers' preferences for the interview location.

IAC nurse(s) and social worker [sample 3] The INSPIRE research team (i.e., Implementation Lead) will give the IAC staff an invitation letter see and a consent form, inviting them to participate in regular meetings with the research team during the feasibility study. The purpose of these meetings will be to regularly explore their perceptions of the IAC with regards to adoption and feasibility of the care model, fidelity, and additional implementation strategies needed.

External collaborators [sample 4] As part of the marketing of the IAC, the IAC manager intends to contact external collaborators (i.e., existing community health and social providers who may have collaborated with the IAC staff for care coordination of a visiting older adult, such as GPs or Spitex Nurses) together with the INSPIRE team, reminding them that the IAC and INSPIRE are working together, and that the INSPIRE team may reach out to them separately. The INSPIRE team will then extract the contact information of collaborating external professionals from the IAC health records of participating older adults. INSPIRE will contact the collaborating professionals and send them a study invitation letter and the NoMAD survey by email (or by paper as an alternative option). The NoMAD aims to assess the IAC implementation processes regarding the collaboration for care coordination. It does not collect any identifying information and only summarized results will be reported.

Study procedures

1. Recruitment feasibility and strategies- external processes: INSPIRE will monitor all IAC promotion activities (e.g., # of letters sent, # of meetings with external groups) and respondents (e.g., # of Hospitals who administer flyers to their staff) at the end of each month during the feasibility study, which will be provided by the IAC.

   Recruitment feasibility and strategies- internal processes: In March 2022, when the feasibility study starts, the IAC administration will provide the INSPIRE research team with summarized administrative data (demographic and IAC use data about all visitors or home appointments) (sample 1A). As part of regular practice, when an older adult arrives at the IAC (or has an appointment at home), they will be asked to complete the standard client information forms and a IAC health record will be created.
2. If the individual is eligible (e.g., home-based older adult aged 64+ with a IAC health record; see criteria for Sample 1B), the IAC nurse will invite them to participate in the INSPIRE Feasibility Study. The IAC nurse will provide the original invitation to the study, while the INSPIRE research team will explain the study, the consent form and conduct the data collection. Proxy consent will be asked for if indicated by the IAC Nurse. Participation in this portion of the feasibility study entails completing an informed consent form and allowing the INSPIRE research team to extract data from their IAC health record to assess fidelity (based on the assessments conducted) and capture variables which describe the sample. The INSPIRE team will review the IAC health records of participating older adults (sample 1B) each week and once at the end of the study to complete the fidelity tool.
3. The informed consent form (described above) also specifies that the individual may be invited to participate in an interview, as the research team will interview a nested sample (sample 1C) of 8-12 older adults. If the older adult is eligible for an interview based on review of their IAC health record (e.g., aged 75+, had a GFI ≥4 and had a CGA), the INSPIRE team will follow-up with the older adult to invite them for the interview. The interview will be approximately 45 minutes and will take place in the IAC or the older adult's home within two-weeks after their second appointment, to gather their perceptions of the care model.
4. At the end of the interview, if an informal caregiver attended the appointment with the older adult, the older adult will be asked if we could invite the informal caregiver for an interview as well (to understand if the informal caregiver perceives the IAC care model to be acceptable and feasible, and if they identify any barriers/facilitators for the older adults' participation in the care model). The INSPIRE team will then reach out to the informal caregiver to provide the study information and consent.

   If a proxy has provided consent for the health record review but not for the interview (or if the older adult does not want to complete an interview), the proxy will still be invited to complete the interview designed for informal caregivers.
5. External providers who are identified in the IAC health records and collaborate with the IAC will also be asked to complete one questionnaire, the NoMAD, at the end of the feasibility study, via an email link to the survey or alternatively in-paper (according to preferences).
6. Throughout the feasibility study, regular meetings will be held with the IAC staff, and one consensus meeting will be held with IAC staff at the end of the feasibility study.
7. All data related to the feasibility study will be collected within 2-3 months. Therefore, data collection will end at the latest by May 31st, 2022.

Data collection or extraction:

1. Recruitment feasibility data

   * External processes data: At the end of each month during the study, INSPIRE will monitor all IAC promotion activities and respondents (provided by the IAC)
   * Internal processes data: The INSPIRE team will capture data provided by the IAC administration at the end of each week, or a mutually agreed time
   * Data will be saved on the research drive of the Institute of Nursing Science
2. IAC health records (of study participants only)

   * A member from the research team will visit the IAC weekly to extract sample characteristics and fidelity data ("39A - Fidelity tool"), using Case Report Forms programmed in Castor, a secure online server (see 7.1)
   * At the end of the study, IAC health records will be accessed again to check if follow-up occurred within the time frame indicated
3. Interview notes and audio recordings with older adults (and informal caregiver, if possible)

   * Conducted within two-weeks of their second appointment
   * Interview notes will be hand-written and scanned into Castor
   * Audio recordings and paper-based notes will be saved in a locked cabinet in the Institute of Nursing Science
4. Meeting logs and audio recordings of meetings with IAC Nurse(s) and social worker

   * Regular meetings will be held
   * Meeting logs will be hand-written and scanned into Castor
   * Audio recordings and paper-based notes will be saved in a locked cabinet in the Institute of Nursing Science
5. NoMAD questionnaire for collaborating health and social care providers

   * Administered towards the end of the study via email through a LimeSurvey link
   * Results will be stored in LimeSurvey, downloaded and saved on the research drive of the Institute of Nursing Science
   * If paper-based survey requested, sent via paper and results will be directly entered into LimeSurvey by INSPIRE research team. Paper-based copy will be stored in a locked cabinet of the Institute of Nursing Science.

Statistical analysis plan Sample size

1. All visitors to the IAC will be included in the assessment of IAC use (1A)
2. All eligible older adults who have a IAC health record created during this time will be invited to participate in the study for review of their IAC health record (1B). While it is currently not possible to provide a precise estimate of the number of visitors to this new center, we estimated a maximum of 18 older adults, estimating 1-2 older adults who visit the IAC each week over a period of 2-2.5 months that will be willing to participate in the study.
3. As we will interview a nested sample (1C), we estimated the sample size for the interviews to be approximately 8-12 older adults. Because analysis will be occurring in parallel with data collection, we estimate information power could likely be achieved in a minimum of 8 interviews (41).
4. We estimate approximately 8-12 informal caregivers (2) [1 per older adult participating in an interview].
5. We estimate 3 IAC staff (3) (i.e., 2 IAC Nurses and 1 Social Worker) to participate in the study.
6. We estimate 18 external collaborators (4), who were involved in the care of the aforementioned 18 older adults, will participate in the study.

Quantitative analysis of feasibility study Descriptive statistics (e.g., mean, median and SD) and frequencies will be calculated and reported to describe the data on recruitment feasibility, participant demographics, study fidelity and survey results.

Qualitative analysis of interviews in the feasibility study Qualitative data from the interviews with participating older adults (as well as their informal caregivers, if possible) will be analyzed using rapid qualitative analysis, as described by Hamilton (42). Two INSPIRE researchers will participate in the interview and take notes on a pre-structured meeting log consistent with the conceptual model domains. A template will be prepared a priori with the main topics to summarize the researchers' meeting notes (42). These notes will be coded, analyzed for themes, and further analyzed using a matrix analysis (42). Interviews will also be audio recorded should further verification or transcription be needed. The main actionable findings will be shared to guide further implementation in real time.

Qualitative analysis of meeting logs in the feasibility study Qualitative data from the meeting logs with the IAC nurse(s) and social worker will be analyzed using rapid qualitative analysis (42), following a similar procedure as described above.

Handling of missing data Missing data will be documented and patterns analyzed. Quality measures

Data Storage:

* Some study data (i.e., fidelity data and information from the IAC health record; demographic information; the researchers' scanned interview notes; the researchers' scanned meeting logs with IAC staff) will be entered/uploaded into CASTOR EDC (Electronic Data Capture), which is a secure online server; it is protected from unauthorized access and access to the database is only possible with personal access data. This data will be double checked by a second individual from the research team (i.e., a PhD student or a Research Assistant/Master's student).
* Other electronic data files (i.e., IAC external and internal processes data in Excel; scanned PDFs of the researchers' interview notes; the IAC staff meeting logs), and the generated excel sheets containing survey results from LimeSurvey (note: LimeSurvey server located in Germany, where full EU GDPR compliance is guaranteed) will be stored on the secure server of the Institute of Nursing Science, where 4 hourly back-ups occur and are mirrored in two different locations and access is controlled by the Active Directory of the University of Basel, which prevents misuse.
* The recordings of the interviews with older adults and informal caregivers, and the audio recordings of the meetings with IAC staff will be securely stored in a locked cabinet at the Institute of Nursing Science, which only two members of the research team will have access (i.e., the Implementation Lead and Academic Lead). The recordings will be saved for a period of 10 years and destroyed thereafter. The paper-based files of the interview notes, the IAC staff meeting notes, and any of the NoMAD questionnaire will also be stored in a locked cabinet at the Institute of Nursing Science.
* For quality assurance, the Ethics Committee may visit the research sites. Direct access to the source data and all study related files is granted on such occasions provided that all involved parties keep the participant data strictly confidential.

Data recording and source data

Data sources:

1. Recruitment feasibility data:

   1. IAC external processes data will be provided by the IAC administration and entered in an Excel file by the INSPIRE research team
   2. IAC internal processes (i.e., IAC use data and demographics): the IAC administrative staff will provide this administrative data to the INSPIRE research team who will enter it into an Excel file
2. IAC health records: the research team will use an electronic case report form (eCRF) for each enrolled older adult in Castor. The older adult will be assigned a unique code (e.g., location - gender - number; "LEIMM1"), to ensure the data is pseudonymized. The first section of the eCRF will include the relevant health-related information to report participant characteristics. The second section of the eCRF will include the fidelity data, based on a review of the IAC health record to document the completed assessments and processes. The eCRF will be filled in by 1 or 2 INSPIRE research team member(s) (i.e., the Implementation Lead or a Research Assistant).
3. Older adult interviews: the researchers' interview notes will be written by hand, scanned and uploaded as an attachment to the eCRF. There will be no identifiable information on the interview notes and only the unique code will be used. If an older adults' informal caregiver also participates in the interview, the written notes will be uploaded as an attachment in the eCRF. The interviews will also be audio recorded.
4. Meeting logs with IAC staff: One eCRF will be completed for each meeting. The researchers' notes obtained through the meetings with IAC staff will be written by hand, scanned and uploaded as an attachment. Demographic data of the IAC staff, which are collected once, (i.e., years of experience and education) will be typed into the eCRF.
5. Questionnaires of external care professionals: The NoMAD questionnaire will be administered via e-mail using a LimeSurvey link (or alternatively available via paper, if requested), and the results stored within LimeSurvey (which have no identifiable information). If any copies are completed by paper, a PhD student or Master's student/research assistant from INSPIRE will enter the survey results directly into LimeSurvey.

For data and query management, monitoring, and reporting, CASTOR EDC will be utilized. This internet-based secure database is developed in agreement with the Good Clinical Practice (GCP) guidelines. The researchers will assure that all data in the course of the study will be entered completely and correctly in this respective database. Access, editing and other corrections in the Castor eCRFs will only be performed by other authorized research team members (i.e., PhD students, Implementation Lead). In case of corrections, the original data entries will be archived in the system and can be made visible. For all data entries and corrections, the date, time of day and person who is performing the entries will be generated automatically. This will ensure that any authorized person who may perform data entries and changes in the eCRF can be identified.

ELIGIBILITY:
Older adults (1A)

All older adults visiting/contacting the Information and Advice Center

Older adults (1B)

Inclusion criteria:

Aged 64 years or older (as this is the statutory retirement age for women in Switzerland and the minimum age of the group we expect to use the Fachstelle services) Living at home German or English-speaking Providing Individual/Proxy Informed Consent (See "3A Informed Consent - Older adult"/"3B Informed Consent -Relative").

Had a Fachstelle health record created

Exclusion criteria:

Residing in a nursing home or planned permanent admission to a nursing home Receiving end-of-life care

Older adults (1C)

Inclusion criteria:

Aged 75 years or older Living at home Living in the participating care region Leimental English or German-speaking Groningen Frailty Indicator [GFI] ≥4 If the older adult had a CGA by the IAC staff Providing Individual/Proxy Informed Consent (See 3A "Informed Consent - Older adult"/ 3B "Informed Consent -Relative")

Exclusion criteria:

Residing in a nursing home or planned permanent admission to a nursing home Receiving end-of-life care Participation in another study with health-related interventions within the 30 days preceding or during the present study GFI < 4 If the older adult did not have a CGA by the IAC staff

Informal caregivers (2)

Inclusion criteria:

Individuals who attended a IAC appointment (in the center or at home) with a participating older adult.

The older adult must agree for the INSPIRE research team to contact the informal caregiver.

Exclusion criteria:

Individuals who did not attend a IAC appointment with a participating older adult or who were not present in a home visit by IAC staff (as the interview questions focus on their perception of the IAC's feasibility and acceptability) Any individuals whom the older adult did not agree for the INSPIRE research team to be contacted

IAC nurse and social worker (3)

Inclusion criteria:

• Individuals employed by the IAC BPA Leimental as a Nurse or Social Worker

Exclusion criteria:

• Other individuals employed by the IAC BPA Leimental (e.g., Administration)

External collaborators (4)

Inclusion criteria:

• Individual health or social care providers who are indicated in the IAC health record as having worked together with the IAC nurse(s) or social worker in the care coordination of a participating older adult

Exclusion criteria:

• Individual health or social care providers who have not contributed to the coordination of care with the IAC staff for a participating older adult

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The groups will be selected from:
  * Residents of the care region of Leimental in Canton Basel-Landschaft in Switzerland: Older adults (1A), Older adults (1B), Older adults (1C), Informal caregivers (2) an
  * Information and Advice Center of the care region of Leimental: nurse and social worker (3)
  * Community (care region of Leimental): External collaborators (4)
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
To assess the adoption of the integrated care model at the IAC, and explore perceptions of IAC staff towards the implemented care model, and if adaptations are needed to the care model or the implementation strategies. | 2 months
  - Adoption is defined as the intention, initial decision, or action to try to employ a new intervention. Adoption will be qualitatively determined during the study through the regular meetings with the IAC Nurse(s) and Social Worker ([sample 3]. These regular meetings will be led by the INSPIRE research team (e.g., Implementation Lead).
To assess the acceptability of the integrated care model at the IAC, and explore perceptions of older adults and their caregivers, IAC staff towards the implemented care model. | 2 months
  - Acceptability is defined as the perception among stakeholders that the intervention is agreeable (31). Acceptability will be captured qualitatively through regular meetings with the IAC Nurse(s) and Social worker (sample 3) as well as through interviews with a nested sample of older adults (e.g., aged 75+, Groningen Frailty Indicator [GFI] score ≥4, received a CGA; see sample 1C) and their informal caregiver (sample 2; e.g., spouse, family member or neighbour), when possible.
To assess the feasibility of the integrated care model at the IAC, and explore perceptions of older adults and their caregivers, and IAC staff towards the implemented care model | 2 months
  - Feasibility is defined as the perception among participating care providers that the intervention is feasible (31). Feasibility will be assessed for recruitment (e.g., referral to the IAC) and aspects of the care model (i.e., screening, CGA, creation of a care plan and collaboration to coordinate care, and follow-up). Feasibility will be captured qualitatively in this study through a) the regular meetings with the IAC staff (sample 3) and b) the interviews with a nested sample of participating older adults (sample 1C) and informal caregivers (sample 2), when possible. A final consensus meeting will be held at the end of the study with the INSPIRE research team, the Head of the IAC and the IAC Nurse(s) and Social Worker to confirm whether the care model is indeed "feasible" and we are ready to move into the effectiveness study.
To assess the fidelity of the integrated care model at the IAC, and explore perceptions of the IAC staff towards the implemented care model, and if adaptations are needed to the care model or the implementation strategies. | 2 months
  - Fidelity is defined as the degree to which the intervention is implemented as it was designed in the original protocol. Fidelity will be quantitatively measured in this study phase by reviewing participating older adults' IAC health records (see sample 1B; e.g., aged 64+, living at home, have a IAC health record) to primarily determine if the care model components (i.e., screening, comprehensive geriatric assessment [CGA], care coordination and individualized care plan, and follow-up were delivered as intended. Fidelity will also be explored qualitatively in the regular meetings with the IAC staff (sample 3).
To explore implementation processes related to collaboration between IAC staff and external health and social care professionals when coordinating care for an older adult | 2 months
  - The Normalization MeAsure Development questionnaire (NoMAD) will be sent to external health and social care providers who have collaborated with the IAC staff for coordination of care of a participating older adult. It is a three-part (A, B, C), 23-item survey. Part A (2-items) asks about their role and job category; in part B, two general questions about the intervention are rated with a response scale of 0-10 (0=not at all, 5=somewhat, 10=completely); and part C (19-items) is in the format of a 5-point Likert scale to indicate level of agreement (1=strongly agree, 3=neutral, 5=strongly disagree). There are four constructs assessed in Part C which are related to the Normalization Process Theory, being: a) coherence (4-items), b) cognitive participation (4-items), c) collective action (7-items; 1 of which we removed due to context), and d) reflexive monitoring (5-items). The NoMAD has a reliability of α = 0.89 for the 20 items and has been cited in many research studies

SECONDARY OUTCOMES:
To assess feasibility of recruitment to the Fachstelle and evaluate recruitment strategies | 2 months
  External processes: monitoring outreach strategies used to promote the IAC to older adults (e.g., letters, brochures) and to sources who could refer/recommend the IAC to older adults (e.g., in-person meetings with Hospitals or Spitex) as well as respondents to the outreach strategies (e.g., # of Hospitals who administer flyers to their staff).
  Internal processes: summarized information related to IAC use of all visitors/home appointments (sample 1A - see Table 2 for criteria), including:
  * number of visitors/home appointment users
  * sociodemographic data of all visitors/home appointments users: age, gender, municipality of residence
  * reason for their appointment/contacting the IAC and referral source (i.e., how they heard about the IAC, and/or the organization which referred them)
  * type of service received by visitors/IAC users: a) health promotion and prevention; b) a full CGA; c) a brief assessment to confirm whether a nursing home referral is warranted; or d) other

OTHER OUTCOMES:
Individual characteristics to describe the sample of consenting older adults (sample 1B) using the IAC services | at baseline: 1 week after enrollment
  * Demographic data: age, gender, and living situation
  * Geriatric risk profile: using the Groningen Frailty Indicator (GFI) where a score of ≥4 represents moderate to severe frailty.
  * Other information to be extracted from the health record of each participant: cognition, depressive symptoms, multimorbidity, nutritional status, and fall history

CONTACTS AND LOCATIONS:
Overall Officials: Sabina M De Geest, Prof. Dr., Principal Investigator — Institute of Nursing Science, University of Basel
Locations (1):
- Fachstelle BPA Leimental (Information and Advice Center of Leimental), Oberwil, Basel-Landschaft, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All data collected in this project will be archived following strictly the current Swiss legal requirements for data protection and will be performed according to the Ordinance HRO Art. 5. Identifying health related data are stored for 10 years after publication of the research project. The delinked study data may be stored longer to answer new research questions, such as in the case of comparative research with national and international groups. The audio recordings will be will be saved for a period of 10 years and destroyed thereafter. At the end of the project, anonymous INSPIRE feasibility study data will be deposited in an appropriate data depository (e.g., Zenodo), as per funding requirements.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will be available at the end of the INSPIRE Project (2024)

REFERENCES:
- [Background] Rechel B, Grundy E, Robine JM, Cylus J, Mackenbach JP, Knai C, McKee M. Ageing in the European Union. Lancet. 2013 Apr 13;381(9874):1312-22. doi: 10.1016/S0140-6736(12)62087-X. Epub 2013 Mar 27. PMID 23541057
- [Background] Donovan NJ, Blazer D. Social Isolation and Loneliness in Older Adults: Review and Commentary of a National Academies Report. Am J Geriatr Psychiatry. 2020 Dec;28(12):1233-1244. doi: 10.1016/j.jagp.2020.08.005. Epub 2020 Aug 19. PMID 32919873
- [Background] Wiles JL, Leibing A, Guberman N, Reeve J, Allen RE. The meaning of "aging in place" to older people. Gerontologist. 2012 Jun;52(3):357-66. doi: 10.1093/geront/gnr098. Epub 2011 Oct 7. PMID 21983126
- [Background] Fuller-Thomson E, Yu B, Nuru-Jeter A, Guralnik JM, Minkler M. Basic ADL disability and functional limitation rates among older AMERICANS from 2000-2005: the end of the decline? J Gerontol A Biol Sci Med Sci. 2009 Dec;64(12):1333-6. doi: 10.1093/gerona/glp130. Epub 2009 Sep 1. PMID 19723771
- [Background] Abdi S, Spann A, Borilovic J, de Witte L, Hawley M. Understanding the care and support needs of older people: a scoping review and categorisation using the WHO international classification of functioning, disability and health framework (ICF). BMC Geriatr. 2019 Jul 22;19(1):195. doi: 10.1186/s12877-019-1189-9. PMID 31331279
- [Background] Parry C, Min SJ, Chugh A, Chalmers S, Coleman EA. Further application of the care transitions intervention: results of a randomized controlled trial conducted in a fee-for-service setting. Home Health Care Serv Q. 2009;28(2-3):84-99. doi: 10.1080/01621420903155924. PMID 20182958
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Leijten FRM, Struckmann V, van Ginneken E, Czypionka T, Kraus M, Reiss M, Tsiachristas A, Boland M, de Bont A, Bal R, Busse R, Rutten-van Molken M; SELFIE consortium. The SELFIE framework for integrated care for multi-morbidity: Development and description. Health Policy. 2018 Jan;122(1):12-22. doi: 10.1016/j.healthpol.2017.06.002. Epub 2017 Jun 20. PMID 28668222
- [Background] Deschodt M, Laurent G, Cornelissen L, Yip O, Zuniga F, Denhaerynck K, Briel M, Karabegovic A, De Geest S; INSPIRE consortium. Core components and impact of nurse-led integrated care models for home-dwelling older people: A systematic review and meta-analysis. Int J Nurs Stud. 2020 May;105:103552. doi: 10.1016/j.ijnurstu.2020.103552. Epub 2020 Feb 29. PMID 32200100
- [Background] Hopman P, de Bruin SR, Forjaz MJ, Rodriguez-Blazquez C, Tonnara G, Lemmens LC, Onder G, Baan CA, Rijken M. Effectiveness of comprehensive care programs for patients with multiple chronic conditions or frailty: A systematic literature review. Health Policy. 2016 Jul;120(7):818-32. doi: 10.1016/j.healthpol.2016.04.002. Epub 2016 Apr 11. PMID 27114104
- [Background] Looman WM, Huijsman R, Fabbricotti IN. The (cost-)effectiveness of preventive, integrated care for community-dwelling frail older people: A systematic review. Health Soc Care Community. 2019 Jan;27(1):1-30. doi: 10.1111/hsc.12571. Epub 2018 Apr 17. PMID 29667259
- [Background] Yip O, Huber E, Stenz S, Zullig LL, Zeller A, De Geest SM, Deschodt M; INSPIRE consortium. A Contextual Analysis and Logic Model for Integrated Care for Frail Older Adults Living at Home: The INSPIRE Project. Int J Integr Care. 2021 Apr 23;21(2):9. doi: 10.5334/ijic.5607. PMID 33976598
- [Background] Smit LC, Schuurmans MJ, Blom JW, Fabbricotti IN, Jansen APD, Kempen GIJM, Koopmans R, Looman WM, Melis RJF, Metzelthin SF, Moll van Charante EP, Muntinga ME, Ruikes FGH, Spoorenberg SLW, Suijker JJ, Wynia K, Gussekloo J, De Wit NJ, Bleijenberg N. Unravelling complex primary-care programs to maintain independent living in older people: a systematic overview. J Clin Epidemiol. 2018 Apr;96:110-119. doi: 10.1016/j.jclinepi.2017.12.013. Epub 2017 Dec 28. PMID 29289764
- [Background] Peters DH, Adam T, Alonge O, Agyepong IA, Tran N. Implementation research: what it is and how to do it. BMJ. 2013 Nov 20;347:f6753. doi: 10.1136/bmj.f6753. No abstract available. PMID 24259324
- [Background] Neta G, Brownson RC, Chambers DA. Opportunities for Epidemiologists in Implementation Science: A Primer. Am J Epidemiol. 2018 May 1;187(5):899-910. doi: 10.1093/aje/kwx323. PMID 29036569
- [Background] Stewart AL, Napoles AM, Piawah S, Santoyo-Olsson J, Teresi JA. Guidelines for Evaluating the Feasibility of Recruitment in Pilot Studies of Diverse Populations: An Overlooked but Important Component. Ethn Dis. 2020 Nov 19;30(Suppl 2):745-754. doi: 10.18865/ed.30.S2.745. eCollection 2020. PMID 33250621
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Finch TL, Girling M, May CR, Mair FS, Murray E, Treweek S, McColl E, Steen IN, Cook C, Vernazza CR, Mackintosh N, Sharma S, Barbery G, Steele J, Rapley T. Improving the normalization of complex interventions: part 2 - validation of the NoMAD instrument for assessing implementation work based on normalization process theory (NPT). BMC Med Res Methodol. 2018 Nov 15;18(1):135. doi: 10.1186/s12874-018-0591-x. PMID 30442094
- [Background] Steverink N, Slaets JPJ, Schuurmans H, van Lis M. Measuring frailty: Developing and testing the GFI (Groningen frailty indicator). Gerontologist. 2001 Oct;41:236-7.
- [Background] Peters LL, Boter H, Buskens E, Slaets JP. Measurement properties of the Groningen Frailty Indicator in home-dwelling and institutionalized elderly people. J Am Med Dir Assoc. 2012 Jul;13(6):546-51. doi: 10.1016/j.jamda.2012.04.007. Epub 2012 May 12. PMID 22579590
- [Background] Integrated care for older people (ICOPE): Guidance for person-centred assessment and pathways in primary care. Geneva: World Health Organization; 2019 (WHO/FWC/ALC/19.1). Licence: CC BY-NC-SA 3.0 I
- [Background] Tsoi KK, Chan JY, Hirai HW, Wong SY, Kwok TC. Cognitive Tests to Detect Dementia: A Systematic Review and Meta-analysis. JAMA Intern Med. 2015 Sep;175(9):1450-8. doi: 10.1001/jamainternmed.2015.2152. PMID 26052687
- [Background] Rubenstein LZ, Harker JO, Salva A, Guigoz Y, Vellas B. Screening for undernutrition in geriatric practice: developing the short-form mini-nutritional assessment (MNA-SF). J Gerontol A Biol Sci Med Sci. 2001 Jun;56(6):M366-72. doi: 10.1093/gerona/56.6.m366. PMID 11382797
- [Background] Lilamand M, Kelaiditi E, Cesari M, Raynaud-Simon A, Ghisolfi A, Guyonnet S, Vellas B, van Kan GA; Toulouse Frailty Platform Team. Validation of the Mini Nutritional Assessment-Short Form in a Population of Frail Elders without Disability. Analysis of the Toulouse Frailty Platform Population in 2013. J Nutr Health Aging. 2015 May;19(5):570-4. doi: 10.1007/s12603-015-0457-4. PMID 25923488
- [Background] Panel on Prevention of Falls in Older Persons, American Geriatrics Society and British Geriatrics Society. Summary of the Updated American Geriatrics Society/British Geriatrics Society clinical practice guideline for prevention of falls in older persons. J Am Geriatr Soc. 2011 Jan;59(1):148-57. doi: 10.1111/j.1532-5415.2010.03234.x. PMID 21226685
- [Background] Malterud K, Siersma VD, Guassora AD. Sample Size in Qualitative Interview Studies: Guided by Information Power. Qual Health Res. 2016 Nov;26(13):1753-1760. doi: 10.1177/1049732315617444. Epub 2016 Jul 10. PMID 26613970
- [Derived] Yip O, Mendieta MJ, Zullig LL, Zeller A, De Geest S, Deschodt M, Siqeca F, Zuniga F, Briel M, Schwenkglenks M, Quinto C, Dhaini S. Protocol for a mixed methods feasibility and implementation study of a community-based integrated care model for home-dwelling older adults: The INSPIRE project. PLoS One. 2022 Dec 21;17(12):e0278767. doi: 10.1371/journal.pone.0278767. eCollection 2022. PMID 36542596
- See also: official website of the INSPIRE Project — https://inspire-bl.unibas.ch/